CLINICAL TRIAL: NCT05183282
Title: The Effectiveness, Safety, and Tolerability of the Nictavi Tarsus Patch in Managing Lagophthalmos in Children and Adolescents
Brief Title: Nictavi Tarsus Patch for Managing Lagophthalmos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angeline Nguyen (Other)
Responsible Party: Sponsor-Investigator, Angeline Nguyen, Assistant Professor of Clinical Ophthalmology, Children's Hospital Los Angeles
Organization: Children's Hospital Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CHLA-21-00354
Record Dates: First submitted 2021-12-07; First posted 2022-01-10 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Lagophthalmos
MeSH Terms: conditions — Lagophthalmos

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Tarsus Patch Group (Experimental): All subjects will receive the Tarsus Patch to be worn and evaluated by the investigator in the clinic and to also be worn at home for 3 nights.
  Interventions: Device: Tarsus Patch

INTERVENTIONS:
Device: Tarsus Patch — The Tarsus Patch is a flexible adhesive device that is applied to the closed upper eyelid and conforms to the curvature of the eyelid to help keep the eyelid in a closed position.
  Other Names: Nictavi Tarsus Patch

SUMMARY:
Lagophthalmos is the inability to completely close the eyelids, which can be caused by conditions such as facial nerve dysfunction and eyelid scarring. Lagophthalmos causes evaporation of the tears, which in turn can lead to damage to the eye and permanent vision loss. Surgical interventions such as tarsorrhaphy or gold/platinum weight implantation can improve lagophthalmos, but these are invasive procedures that are not easily reversible. Temporary methods for treating lagophthalmos are also available, such as the use of medical tape or commercial eyelid closure devices. In the investigators' clinical experience, however, these methods are not well-tolerated by patients due to discomfort, especially due to the device sticking to the eyelashes. As a result, patients are at greater risk of non-compliance and subsequently experiencing ocular complications.

The Nictavi Tarsus Patch is a new medical device that uses a flexible material that conforms to the upper eyelid curvature while maintaining sufficient rigidity to keep the upper eyelid in a closed position. It also is designed to be placed above the eyelash line, which allows for enhanced comfort. There has been no study to date evaluating the Tarsus Patch for its effectiveness, safety, or tolerability.

The purpose of this study is to determine the effectiveness, safety, and tolerability of the Tarsus Patch in managing lagophthalmos in children and adolescents overnight. The investigators hypothesize that there will be a significant improvement in eyelid closure when using the Tarsus Patch when compared to not using any device and that over 90% of subjects will achieve complete eyelid closure with its use. The investigators also hypothesize there will be no complications related to the use of the Tarsus Patch, and that it will be considered by patients and parents to be comfortable, easy to use, and, overall, preferable to other available methods of nocturnal eyelid closure.

DETAILED DESCRIPTION:
The investigators plan to recruit 20 children and adolescents (ages 0 to 17 years, inclusive) from the Children's Hospital Los Angeles (CHLA) ophthalmology clinics who have lagophthalmos affecting one or both eyes and have been recommended to use medical tape or other eyelid closure device to help keep their eyelids closed. The aims are to 1) objectively measure the improvement in lagophthalmos from baseline while using the Tarsus Patch, and 2) evaluate patients' and parents' experience with survey questions related to complications, comfort, ease of use, and preference for using the about the Tarsus Patch.

PROCEDURES INVOLVED

* Study visit (Day 1 of study, 60 minute commitment):

  * At the study visit, informed consent will be obtained by the study coordinator or investigator.
  * Once consent is obtained, the enrolled subject then undergoes an ophthalmic history and examination, including dilated examination if deemed necessary for their usual ophthalmic care. The history will include usual questions asked at a follow-up visit about ocular health and will also include details about how often, in which eye, and with what method they close their eyelids at night.
  * The examination will include standard measures of vision, ocular surface health, and eyelid position and function.
  * If the subject has unilateral lagophthalmos, then the involved eye will be designated as the study eye. If the subject has bilateral lagophthalmos, then the eye with more severe lagophthalmos will be designated as the study eye.
  * The parent will receive an explanation about the procedures of the study.
  * The study investigator will choose which Tarsus Patch size (pediatric or adult) will fit best on the child's eyelid. With the proper size, the parent will then be shown how to properly place the Tarsus Patch on the study eye, and questions will be answered about how to properly place the patch on the eye.
  * The parent will then be given the following items to take home: 6 patches (this includes a few extra patches in case they are needed), and a copy of the study consent form including email and phone number to reach the study team should they have any questions
  * To minimize risk, the parent will be informed that if the subject has any discomfort with an of the study protocols, they should stop the use of the Patch call the study team to discuss how to address the issue.
* At home portion (Day 1-3 of study):

  - Each night for 3 nights, the parent should place a new Tarsus Patch on the subject's study eye and then place a ½ cm strip of ophthalmic ointment or gel into the study eye. The parent should then help remove the patch the next morning and throw it away.
* Phone survey (Day 4):

  * A study investigator will call the parents to have them respond to the Parent Survey over the phone in the absence of the study subject.
  * If the subject is 10 years of age or older and cognitively able to answer the survey questions, then they will be asked to answer the Subject Survey over the phone with the help of the parent.

ELIGIBILITY:
Inclusion Criteria:

* Patient subjects:

  * Between 0 and 17 years old (inclusive)
  * Diagnosis of unilateral or bilateral lagophthalmos based upon an eye examination since Jan 1, 2019
  * Previously recommended to use an eyelid closure method (such as using medical tape, steristrips, moisture chambers, temporary tarsorrhaphy, etc).
  * English-speaking
  * Able to participate in an age-appropriate manner for the eye examination
* Parent subjects:

  * 18 years or older
  * English-speaking

Exclusion Criteria:

* Patient subjects:

  * Presence of corneal abrasion or corneal ulcer on the study eye
  * Active use of bandage contact lens in the study eye
  * Active dermatitis affecting the eyelids
  * Inability to tolerate the Tarsus Patch in clinic
  * Inability for complete mechanical closure of the eyelid by any means
  * Allergy to adhesive
* Parent subjects:

  * Prisoners

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Lagophthalmos in "eyes closed" position | This measurement is taken on day 1 during the study visit in clinic, which will take about 1 minute.
  While the subject is being asked to close their eyes like they're going to sleep, the amount of lagophthalmos (the distance between the upper and lower eyelid) will be measured in millimeters. This measurement will be taken both while the subject is wearing the Tarsus Patch on the study eye and while the subject is not wearing the Tarsus Patch on the study eye. The difference in average lagophthalmos between when the Tarsus Patch is on versus off will be analyzed by paired t-test.

SECONDARY OUTCOMES:
Interpalpebral fissure distance in upgaze | This measurement is taken on day 1 during the study visit in clinic, which will take about 1 minute.
  While the subject is being asked to look upwards, the interpalpebral fissure distance (distance between the upper and lower eyelid) will be measured in millimeters. This measurement will be taken both while the subject is wearing the Tarsus Patch on the study eye and while the subject is not wearing the Tarsus Patch on the study eye. The difference in average interpalpebral fissure distance between when the Tarsus Patch is on versus off will be analyzed by paired t-test.
Parental and subjects' subjective experience using the Tarsus Patch | These surveys will be administered by phone on day 4, which is after the last day the subject wears the Tarsus Patch at home. The survey should take about 3 minutes per person.
  The parent and subject (if 10 years of age or older) will be asked a series of likert-style questions that assess the comfort, ease of use, and preferability of the Tarsus Patch.
Parental report of safety while using the Tarsus Patch | The parental survey will be administered by phone on day 4, which is after the last day the subject wears the Tarsus Patch at home. The survey should take about 3 minutes per person.
  Parents will be asked to report and elaborate during their survey if they felt that there were any complications or adverse effects related to using the patch.

CONTACTS AND LOCATIONS:
Overall Officials: Angeline M Nguyen, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Latkany RL, Lock B, Speaker M. Nocturnal lagophthalmos: an overview and classification. Ocul Surf. 2006 Jan;4(1):44-53. doi: 10.1016/s1542-0124(12)70263-x. PMID 16671223
- [Background] Masoudi Alavi N, Sharifitabar Z, Shaeri M, Adib Hajbaghery M. An audit of eye dryness and corneal abrasion in ICU patients in Iran. Nurs Crit Care. 2014 Mar;19(2):73-7. doi: 10.1111/nicc.12052. Epub 2013 Oct 16. PMID 24131554